CLINICAL TRIAL: NCT05678907
Title: Predictive Value of the DD4 Questionnaire on Depressive Relapse After Hospitalization
Acronym: PRADESH
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2022-06-054
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Depressive Episode

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal, single-center observational study of data from the medical records of patients hospitalized after a characterized depressive episode and reviewed three months after hospital discharge, as part of a normally scheduled evaluation.

DETAILED DESCRIPTION:
Patients in the study were hospitalized following a characterized depressive episode. The study is based on a review of these patients' medical records and data from the three-month assessment. No additional assessments are planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older, having been informed of the research
* Patient hospitalized at the Auzon Clinic for a characterized depressive episodé (isolated episode or recurrent depressive disorder)
* Discharged from hospitalization
* Considered in remission (total or partial) and with a MADRS score < 20

Exclusion Criteria:

* Patient hospitalized for < 15 days
* Patient with bipolar depression
* Patient with a psychotic disorder
* Patient using narcotics with a "moderate to severe" severity
* Patient previously included in this study
* Patient under court protection, guardianship or curatorship
* Patient unablé to respond correctly to a depression self-assessment questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for a characterized depressive episode and considered in remission at discharge.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Depressive episode relapse | Month 3
  Relapse within three months of hospitalization

SECONDARY OUTCOMES:
Psychic symptoms of depression | Month 3
  The Multidimensional Self-Questionnaire for Depression Assessment DD4 (Ducher's Depression Scale) is presented in the form of four modules.
  Each module consists of 15 identical questions (I feel sad, I suffer morally...).
  The formulation of the questions allows for evaluation from 0 to 4 in different dimensions:
  DD4 A: Global Evaluation (not at all true, a little true, rather true, very true, completely true) DD4 F: Frequency Evaluation (never, sometimes, often, very often, permanently) DD4 I: Intensity Evaluation (not at all, slightly, fairly, a lot, enormously) DD4 M: Maximal Evaluation (uses the criteria of the global evaluation, but during the moments when the patient feels the saddest or most depressed). An additional question asks about the frequency of these periods (never, sometimes, often, very often, permanently).
Depressive symptomology | Month 3
  Measured with the Montgomery and Asberg (MADRS) scale

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Auzon, La Roche-Blanche, France

IPD SHARING:
Plan to Share IPD: No